CLINICAL TRIAL: NCT05214287
Title: An N-of-1 Double-blind Randomized Phase 1 Trial of the Safety and Feasibility of (Intermittent) Hypoxia Therapy in Parkinson's Disease (TALISMAN)
Brief Title: Multiple N-of-1 Trials of (Intermittent) Hypoxia Therapy in Parkinson's Disease
Acronym: TALISMAN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 112203; NL.77891.091.21 (Other: ToetsingOnline.nl); 2021-005480-41 (EudraCT Number); 2021-12410 (Other: Medical Ethics Research Committee East-Netherlands)
Record Dates: First submitted 2021-12-28; First posted 2022-01-28 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease; Effect of Drug
Keywords: Parkinson's disease; Treatment; Intermittent hypoxia therapy; IHT; Disease-modifying treatment; Symptomatic therapy; Neurodegenerative Diseases; Synucleinopathies; Oxygen Deficiency; Hypoxia, Brain; Movement Disorders
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases; Synucleinopathies; Hypoxia; Hypoxia, Brain; Movement Disorders | interventions — nitrox

STUDY DESIGN:
Intervention Model Description: The investigators will deploy an N-of-1 trial design (also known as single participant cross-over trial) in which multiple treatment pairs of active treatment and placebo are offered to an individual participant in a randomized, double-blind fashion. In an N-of-1 trial, random variation within the treatment effect at the individual level can be better accounted for and methodological power is optimized due to repeated treatment-pairs and the fact that the individual participant acts as their own control. Thanks to this design, in which each treatment-pair should be exchangeable in time, N-of-1 trials are especially suitable to investigate treatments in chronic, symptomatic conditions, where period effects (i.e. changes in disease state) and carry over effects (i.e. lingering hypoxia effects) are small. Given the slowly progressive nature of PD with relative stable symptoms, several N-of-1 trials have already been successfully performed to study symptomatic treatments in PD.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The administration and sequence of intervention(s) will not be disclosed to the participant. However, due to the n-of-1 design, all participants will be exposed to all treatment modalities as well as the control condition arm, which makes concealed allocation not applicable other than the unconcealed intervention sequence. The investigators will assess success of masking by asking a participant in what sequence the different treatments were probably administered.
  For safety and monitoring purposes, the intervention is not blinded for the lab technician, who will administer and monitor the intervention.
  All outcomes will be assessed directly before and after the stimulus by an independent and blinded assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Intermittent with 5x5-minutes, FiO2 0.163 (Experimental): Delivered intermittently, with FiO2 0.163 and room-air, each 5 minutes, for 5 cycles/session
  Interventions: Drug: Hypoxic Gas Mixture
- Intermittent with 5x5-minutes, FiO2 0.127 or 0.133 (Experimental): Delivered intermittently, with FiO2 0.127 or 0.133 (depending on SaO2 during screening procedure at FiO2 0.127, see study procedures) and room-air, each 5 minutes, for 5 cycles/session
  Interventions: Drug: Hypoxic Gas Mixture
- Continuous for 45 minutes, FiO2 0.163 (Experimental): Delivered via the hypoxicator
  Interventions: Drug: Hypoxic Gas Mixture
- Continuous for 45 minutes, FiO2 0.127 or 0.133 (Experimental): FiO2 0.127 or 0.133 (depending on SaO2 during screening procedure at FiO2 0.127, see study procedures)
  Interventions: Drug: Hypoxic Gas Mixture
- Continuous for 45 minutes, FiO2 0.209 (Placebo Comparator): Delivered via an open three-way valve in the circuitry from hypoxicator to the participant
  Interventions: Drug: Hypoxic Gas Mixture

INTERVENTIONS:
Drug: Hypoxic Gas Mixture — Using a commercially available hypoxicator, varying gas mixtures as described will be administered via a tight-fitting oxygen mask. In the circuitry, a three-way valve is placed that allows for the intermittent administration of hypoxia: the valve either passes the hypoxic mixture from the hypoxicator or room air.
  Other Names: Hypoxicator

SUMMARY:
In recent years, mitochondrial dysfunction and oxidative stress have been implicated in PD pathophysiology. Intermittent hypoxia therapy (IHT) is an upcoming treatment used by elite athletes as well as fragile individuals in clinical settings that works by improving exercise tolerance, neuroplasticity and inducing hypoxic preconditioning (HPC). HPC might improve the oxidative stress response in PD on the long-term. In addition, preclinical evidence suggests beneficial short-term effects such as influence on dopamine and noradrenalin release. Anecdotal evidence indeed suggests that visiting high-altitude areas improves PD symptoms and it is hypothesized that this effect results from decreased oxygen pressure at high altitudes. The safety and feasibility of (intermittent) hypoxia therapy on PD symptoms will be assessed in an exploratory phase I randomized-controlled trial.

DETAILED DESCRIPTION:
Parkinson's disease (PD) currently affects 10 million people worldwide and its prevalence is projected to exponentially rise further in the absence of disease-modifying therapies. A scarcity of symptomatic treatments is available and the mainstay of therapy has been levodopa for over half a century. Although this treatment suffices for many patients in early phases of PD, treatment burden is significant, as are the adverse effects, wearing-off and dyskinesia that develop with disease progression. Therefore, additional treatment modalities are needed.

Preclinical studies have suggested that moderate hypoxia provokes release of survival-enhancing neurotransmitters, such as dopamine release from the substantia nigra. Clinical and preclinical evidence suggests the effects of hypoxia seem especially robust when applied using intermittent hypoxia therapy (IHT) compared to continuous hypoxia. IHT means that hypoxia is present for relatively short periods (i.e. minutes), interspersed with short periods of recovery at normoxia (i.e. sea-level). The precise working mechanism of IHT on the short term remains unclear, but the immediate clinical effects appear to be related to augmented dopamine release from the substantia nigra. Specifically, IHT may improve parkinsonian symptoms via activation of the Hypoxia Inducible Factor 1 (HIF-1) pathway, which in turn activates tyrosine hydroxylase (TH), which is the main rate-limiting enzyme in the production of dopamine. Several studies have demonstrated that HIF-1 stabilization leads to an increase in TH production, and consequently a rise in cellular dopamine content. IHT is a therapy proven safe and effective in a variety of disciplines, including fragile populations such as individuals with chronic obstructive pulmonary disorder (COPD), cardiac morbidity and spinal cord injury. Long-term application of IHT protocols was associated with improved oxidative stress response and adaptive plasticity in the dopaminergic system of rodents, suggesting that in addition to the acute symptomatic effects, repeated exposure to (intermittent) hypoxia might also exert some long-term neuroprotective effects. The general concept behind a possible (long-term) neuroprotective effect of IHT is the phenomenon of hypoxic conditioning: induction of a sub-toxic hypoxic stimulus to improve the (systemic) tolerance of cells and tissues to subsequent more severe stimuli, either in dose or duration. In this way, key adaptive mechanisms are induced that allow maintenance of cellular homeostasis under low-oxygen conditions. Among these adaptive mechanisms, activation of HIF-1 is the most prominent and most extensively described mechanism. Interestingly, IHT protocols also blocked the neurotoxic effect of agents that induce PD in rodents, preventing development of locomotor deficits, again suggesting some neuroprotective effects. Furthermore, circumstantial anecdotal evidence from individuals with PD suggests that ascending to high-altitude areas (e.g. on holidays) improves motor symptoms of PD, which the investigators recently confirmed in a survey conducted in the holiday context (https://doi.org/10.1002/mdc3.13597). The investigators hypothesize that the positive effect of altitude on the symptoms of PD result from decreased oxygen pressure at high altitude, which serves as an acute bodily stressor that releases survival-enhancing neurotransmitters such as dopamine and noradrenaline and might induce neuroprotective mechanisms.

The investigators will assess the potential of IHT in PD by assessing symptomatic effects of intermittent hypoxia therapy in an exploratory phase I trial. Primary objectives are the safety and feasibility of intermittent hypoxia in PD and assessing the responsiveness of subjective and standardized symptom scales to this intervention. This trial will exploit an aggregated N-of-1 approach, which allows testing multiple high-altitude simulation protocols and outcome measures, analysis of the treatment effect in individuals as it can account for random variation for treatment effects in the individual and enhances methodological power due to repeated treatment pairs.

During a screening procedure, participants undergo pulmonary function testing, carbon monoxide diffusion capacity testing and electrocardiography. If no cardiorespiratory abnormalities are demonstrated, individuals undergo a hypoxic intervention with gradually decreasing FiO2 levels from room air to either FiO2 0.127 or an arterial oxygen saturation (SaO2) of 80%, under vital parameter and blood gas monitoring. If a participant reaches FiO2 0.127 without SaO2 <80%, the most intense active interventions will contain that FiO2. If a participant has an SaO2 <80% before FiO2 0.127 is reached but still has an SaO2 of 80% or higher at FiO2 0.133, the most intense active intervention will be FiO2 0.133 instead of 0.127 (see Interventions)

ELIGIBILITY:
Inclusion criteria:

* Informed consent
* Clinical diagnosis of Parkinson's disease by a movement disorder specialized neurologist with Hoehn and Yahr staging 1.5 to 3.
* 15 individuals with self-reported personal experience of positive altitude effect.
* 5 individuals without self-reported personal experience of positive altitude effect.

Exclusion criteria:

* Individuals with diseases leading to restrictive and obstructive pulmonary diseases, pulmonary diffusion deficits, apnea and cardiac output deficits, such as pulmonary fibrosis, COPD, sleep apnea or excessive alcoholic intake, and congestive heart failure respectively.
* Arterial blood gas abnormalities at screening day (as per normal limits)
* Individuals with shortness of breath or other airway or breathing-related inconvenience related to lack of dopaminergic medication will be excluded.
* Inability to comply to intervention in off-medication condition (for example due to extreme discomfort, distress or severe head tremor due to being OFF, i.e. without dopaminergic medication).
* Individuals with unstable dopaminergic medication dose (changes in the last month)
* Individuals likely to start dopaminergic treatment in the next month, also judged by their treating neurologist
* Individuals with active deep brain stimulation
* Individuals unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Nature and number of adverse events | Until 3 days post-intervention
  Actively reported during intervention and passively for up to 3 days after the intervention, adverse events will be collected.
Self-reported dizziness, discomfort and stress on a ten-point scale | Until 3 days post-intervention
  Every 10 minutes up to one hour post-intervention, one time next morning post-intervention, 10-point Likert scale, lower is better.
Blood pressure | Baseline and every 5 mins until 30 mins post-intervention
  Systolic and diastolic blood pressure
Heartrate | Baseline and every 5 mins until 30 mins post-intervention
  Beats/min
Respiratory rate | Baseline and every 5 mins until 30 mins post-intervention
  Breaths/min
Oxygen saturation | Baseline and every 5 mins until 30 mins post-intervention
  Percentage
Feasibility questionnaire | After 1st, 5th, 10th post-intervention test
  17-item scale, scored 1-10, lower is better. Subscores and total score

SECONDARY OUTCOMES:
Participant-selected motor symptom | Directly after, as well as 30 and 60 minutes after the intervention and four times once every hour after that. In addition, these will be measured once every morning (i.e. in OFF) for the next three mornings after the intervention.
  Change from (pre-treatment) baseline in the symptom that improved most during previous positive altitude effect (if applicable), or other symptom of choice. Self-reported severity scores on a Likert-scale. 10-point Likert scale allowing half points. Lower is better.
General impression of PD symptoms | Directly after, as well as 30 and 60 minutes after the intervention and four times once every hour after that. In addition, these will be measured once every morning (i.e. in OFF) for the next three mornings after the intervention.
  Change from (pre-treatment) baseline on 10-point Likert scale allowing half points. Lower is better.
Urge to take dopaminergic medication | Directly after, as well as 30 and 60 minutes after the intervention and four times once every hour after that. In addition, these will be measured once every morning (i.e. in OFF) for the next three mornings after the intervention.
  Change from (pre-treatment) baseline on 10-point Likert scale allowing half points. Lower is better.
Timed Up & Go Test | 30 minutes
  Change from (pre-treatment) baseline in total time and steps. The Timed Up & Go Test is a test that evaluates primarily gait functioning. Lower is better.
MiniBESTest | 30 minutes
  Change from (pre-treatment) baseline in item subscores and total score. The MiniBESTest is a concise balance test. Higher is better.
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III | 30 minutes
  The MDS-UPDRS part III is the gold standard for motor assessment in Parkinson's disease. Change form (pre-treatment) baseline in item subscores and total scores. Lower is better.
Finger tapping | 30 minutes
  Change from (pre-treatment) baseline in number of taps during 10-second trials on both hands, one session each. Finger tapping is considered a measure of bradykinesia. Higher is better.
MDS Non-Motor Symptoms Scale (only items related to stress, fatigue, mood, anxiety, pain) | 30 minutes
  The most important potentially adaptive non-motor symptoms mentioned in this gold standard for non-motor symptom screening are selected. Likert scale 1-10 (allowing half points). Change from (pre-treatment) baseline. Lower is better.
Accelerometry during MDS-UPDRS part III, items on pronation-supination and tremor | 30 minutes
  During the MDS-UPDRS part III, accelerometry allows for quantification of therapeutic effects in addition to the MDS-UPDRS part III. Lower amplitude is better in tremor, higher frequency and rotational power is better in pronation-supination. Change from (pre-treatment) baseline.
Heart Rate Variability (HRV) | 30 minutes
  Average HRV during intervention and post intervention. HRV is a marker of cardiovascular stress. Change form (pre-treatment) baseline. Lower equals more stress.
Modified Purdue pegboard test | 30 minutes
  Change from (pre-treatment) baseline in number of pins per side. The Purdue pegboard test is primarily a measure of bradykinesia, hypokinesia and fine motor skills. Higher is better.

OTHER OUTCOMES:
Serum platelet-derived growth factor receptor β (PDGFRβ) | 60 minutes after intervention
  PDGFRβ is a pericyte-released marker of hypoxia and blood-brain barrier integrity. Change from (pre-treatment) baseline. Higher equals more hypoxic-induced adaptive response
Serum cortisol | Directly after intervention, 30 minutes, 60 minutes
  Cortisol is a molecular marker of systemic stress. Change from (pre-treatment) baseline. Lower equals less stress.
Serum erythropoietin (EPO) | 60 minutes after intervention
  Erythropoietin is a marker of cellular hypoxia. Change from (pre-treatment) baseline. Higher equals more hypoxic-induced adaptive response.

CONTACTS AND LOCATIONS:
Overall Officials: prof. dr. Bastiaan R. Bloem, Principal Investigator — Center of Expertise for Parkinson and Movement Disorders, Radboud university medical center; prof. dr. Dick H.J. Thijssen, Principal Investigator — Department of Integrative Physiology, Radboud university medical center
Locations (1):
- Dpt. of Physiology, Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared with The Michael J. Fox Foundation for Parkinson's Research (the study funder). This data may be kept for storage at a central repository either hosted by The Michael J. Fox Foundation, its collaborators, or consultants and will be kept indefinitely. Anonymized data will be made publically available for the intended use of research in Parkinson's disease as well as other biomedical research studies that may not be related to Parkinson's disease.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be made available within 1.5 years after study completion date.
Access Criteria: Access to and use of data are supervised by the Michael J. Fox Foundation.

REFERENCES:
- [Derived] Janssen Daalen JM, Meinders MJ, Giardina F, Roes KCB, Stunnenberg BC, Mathur S, Ainslie PN, Thijssen DHJ, Bloem BR. Multiple N-of-1 trials to investigate hypoxia therapy in Parkinson's disease: study rationale and protocol. BMC Neurol. 2022 Jul 14;22(1):262. doi: 10.1186/s12883-022-02770-7. PMID 35836147